CLINICAL TRIAL: NCT02371980
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 4, Relapse Prevention Study Evaluating the Efficacy and Safety of Vortioxetine (5, 10 and 20 mg) in Adults With Major Depressive Disorder
Brief Title: Vortioxetine, 5, 10, and 20 mg, Relapse Prevention Study in Adults With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LuAA21004_402; U1111-1161-4956 (Registry Identifier: WHO)
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Results first posted 2020-04-17 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Major Depressive Disorder
Keywords: Drug therapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Open-label: Vortioxetine 10 mg (Experimental): Vortioxetine 10 mg, capsules, orally, once, daily (QD) up to 8 weeks. Participants who achieved response (defined as a ≥50% reduction in Montgomery Asberg Depression Rating Scale (MADRS) total score from Baseline) continued to receive vortioxetine 10 mg, capsules, orally, QD for up to Week 16 (stabilization period) in the Open-label Period.
  Interventions: Drug: Vortioxetine
- Double-blind: Placebo (Placebo Comparator): Following Open-label Period, participants who achieved remission criteria (defined as MADRS total score ≤12 at Weeks 14 and 16) were randomized to receive vortioxetine placebo-matching capsules, orally, QD from Week 17 up to Week 44 in the Double-blind Period.
  Interventions: Drug: Placebo
- Double-blind: Vortioxetine 5 mg (Experimental): Following Open-label Period, participants who achieved remission criteria (defined as MADRS total score ≤12 at Weeks 14 and 16) were randomized to receive vortioxetine 5 mg, capsules, orally, QD from Week 17 up to Week 44 in the Double-blind Period.
  Interventions: Drug: Vortioxetine
- Double-blind: Vortioxetine 10 mg (Experimental): Following Open-label Period, participants who achieved remission criteria (defined as MADRS total score ≤12 at Weeks 14 and 16) were randomized to receive vortioxetine 10 mg, capsules, orally, QD from Week 17 up to Week 44 in the Double-blind Period.
  Interventions: Drug: Vortioxetine
- Double-blind: Vortioxetine 20 mg (Placebo Comparator): Following Open-label Period, participants who achieved remission criteria (defined as MADRS total score ≤12 at Weeks 14 and 16) were randomized to receive vortioxetine 20 mg, capsules, orally, QD from Week 17 up to Week 44 in the Double-blind Period.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Vortioxetine capsules
  Other Names: LuAA21004
  Arms: Double-blind: Vortioxetine 10 mg; Double-blind: Vortioxetine 20 mg; Double-blind: Vortioxetine 5 mg; Open-label: Vortioxetine 10 mg
Drug: Placebo — Vortioxetine placebo-matching capsules
  Arms: Double-blind: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of vortioxetine (5, 10, and 20 mg) versus placebo during the first 28 weeks of the 32-week double-blind treatment period in the prevention of relapse in participants with MDD who responded to acute treatment with vortioxetine 10 mg.

DETAILED DESCRIPTION:
The drug being tested in this study is called vortioxetine. Vortioxetine is being tested for the prevention of relapse in adults with major depressive disorder (MDD) who respond to daily treatment with vortioxetine. This study will look at relapse rates of MDD in people who take vortioxetine.

The study will enroll approximately 1100 participants. All participants will receive vortioxetine 10 mg open-label for the first 16 weeks of the study. Participants who meet the appropriate MDD response criteria from the Week 8 Visit through Week 16 Visit will be eligible for randomization into the double-blind treatment period. Participants will be randomly assigned (by chance, like flipping a coin) to one of the four treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Vortioxetine 5 mg
* Vortioxetine 10 mg
* Vortioxetine 20 mg
* Placebo (dummy inactive pill) - this is a capsule that looks like the study drug but has no active ingredient

All participants will be asked to take one capsule at the same time each day throughout the study.

This multi-center trial will be conducted in the United States. The overall time to participate in this study is up to 55 weeks. Participants will make 19 visits to the clinic, and will be contacted by telephone 4 weeks after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Suffers from recurrent major depressive disorder (MDD) as the primary diagnosis according to Diagnostic & Statistical Manual of Mental Disorders, 4th Edition - Text Revision (DSM-IV-TR) criteria (classification code 296.3x), and the current episode is confirmed by the Mini International Neuropsychiatric Interview (MINI).
4. Reported duration of the current episode is ≥8 weeks and ≤18months.
5. Had at least 2 other major depressive episodes (MDEs) before the current episode.
6. Has a Montgomery-Åsberg Depression Rating Scale (MADRS) total score ≥26 at the Screening and Baseline I visits.
7. Is a man or woman aged 18 to 75 years, inclusive.
8. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from signing of the informed consent throughout the duration of the study and for 30 days after the last dose.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to screening or 5 half-lives prior to screening, whichever is longer.
2. Has previously or is currently participating in this study.
3. Has participated in 2 or more clinical studies in the year prior to screening, or has participated in a clinical trial for a psychiatric condition that is exclusionary per this protocol.
4. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
5. Has one or more of the following:

   1. Any current psychiatric disorder which is the primary focus of treatment other than MDD as defined in the DSM-IV-TR, and assessed by the MINI.
   2. Current or history of: manic or hypomanic episode, schizophrenia or any other psychotic disorder, including schizoaffective disorder, major depression with psychotic features, bipolar depression with psychotic features, obsessive compulsive disorder (OCD), mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR.
   3. Current diagnosis or history of alcohol or other substance abuse or dependence (excluding nicotine or caffeine) as defined in the DSM-IV-TR that has not been in full and sustained remission for at least 3 months from the day of screening (Participant must also have negative urine drug screen at Screening and Baseline I.)
   4. Presence or history of a clinically significant neurological disorder (including epilepsy) as determined by the investigator.
   5. Neurodegenerative disorder (Alzheimer disease, Parkinson disease, multiple sclerosis, Huntington disease, etc).
   6. Any Axis II disorder as defined by DSM-IV-TR that might compromise the study.
6. The current depressive symptoms of the participant are considered by the investigator to have been resistant to 2 adequate antidepressant treatments of at least 6 weeks duration each.
7. Has a history of lack of response to previous adequate treatment with vortioxetine for any MDD episode with adequate treatment considered to be known dose of vortioxetine in the approved recommended dose range for at least 6 weeks duration.
8. Has received electroconvulsive therapy, vagal nerve stimulation, or repetitive transcranial magnetic stimulation within 6 months prior to Screening.
9. Has started receiving formal cognitive or behavioral therapy, systematic psychotherapy within 30 days from screening or plans to initiate such therapy during the study (supportive therapy, marital therapy and bereavement counseling are allowed).
10. Has a significant risk of suicide according to the investigator's clinical judgment or has a score ≥5 on item 10 (suicidal thoughts) of the MADRS or has made a suicide attempt in the previous 6 months.
11. Is required to take excluded medications or it is anticipated that the participant will require treatment with at least 1 of the disallowed concomitant medications during the study.
12. Has a clinically significant unstable illness, for example hepatic impairment or renal insufficiency, or a cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, rheumatologic, immunologic, hematological, infectious, dermatological disorder or metabolic disturbance.

    Note: For the purposes of this protocol fibromyalgia, obstructive sleep apnea, chronic pain diagnosis, and morbid obesity (BMI of > 40) are considered unstable due to the potential impact on assessment of the primary endpoint.
13. Has a known history of or currently has increased intraocular pressure or is at risk of acute narrow-angle glaucoma.
14. Has 1 or more laboratory value outside the normal range, based on the blood or urine samples taken at the Screening Visit, that are considered by the investigator to be clinically significant; or the participant has any of the following values at the Screening Visit:

    1. A serum creatinine value >1.5 times the upper limits of normal (ULN).
    2. A serum total bilirubin value >1.5 xULN.
    3. A serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value >2 xULN.
15. Has glycosylated hemoglobin (HbA1C) ≥7% at screening and no prior diagnosis of diabetes and/or treatment for diabetes. NOTE: Participants with known stable diabetes are not excluded.
16. Has a thyroid stimulating hormone (TSH) value outside the normal range at the Screening Visit that is deemed clinically significant by the investigator. NOTE: Free T4 will be checked if TSH is out of range. If free T4 is abnormal the participant will be excluded.
17. Has clinically significant abnormal vital signs as determined by the investigator.
18. Has an abnormal electrocardiogram (ECG) as determined by the central reader and confirmed as clinically significant by the investigator.
19. Is positive for Hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies, or has a history of human immunodeficiency virus (HIV) infection.
20. Has a disease or takes medication that, in the opinion of the investigator, could interfere with the assessments of safety, tolerability or efficacy.
21. The participant, in the opinion of the investigator, is unlikely to comply with the clinical study protocol or is unsuitable for any reason.
22. Has a history of hypersensitivity or allergies to vortioxetine.
23. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
24. The participant is considered to be treatment resistant, eg, the participant has not responded to adequate monotherapy treatments of at least 6 weeks' duration, or has only responded to combination or augmentation therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1106 (Actual)
Dates: Start 2015-02-10 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (79):
- United States (79):
  - NoesisPharma, Phoenix, Arizona
  - SW Biomedical Research, LLC, Tucson, Arizona
  - CNS Research Science, Inc., Cerritos, California
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Irvine Center for Clinical Research, Inc., Irvine, California
  - Synergy Clinical Research of Escondido, Lemon Grove, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pacific Institute of Medical Research, Los Angeles, California
  - CNRI - Los Angeles, LLC, Pico Rivera, California
  - CNRI - San Diego, LLC, San Diego, California
  - Artemis Institute for Clinical Research, LLC, San Diego, California
  - University of California San Diego Medical Center, San Diego, California
  - Pasadena Research Institute, San Gabriel, California
  - Collaborative Neuroscience Network, LLC, Torrance, California
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - CNS Clinical Research Group, Coral Springs, Florida
  - Gulfcoast Medical Research Center, LLC, Fort Myers, Florida
  - MD Clinical, Hallandale, Florida
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Meridien Research, Maitland, Florida
  - Sarkis Clinical Trials - Parent, Ocala, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Janice L. Miller, M.D., PA d/b/a Janus Center for Psychiatric Reseach, West Palm Beach, Florida
  - Radiant Research, Inc., Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Alexian Brothers Center for Psychiatric Research, Arlington Heights, Illinois
  - Rush St Lukes Presbyterian Medical Center, Chicago, Illinois
  - Capstone Clinical Research, Inc., Libertyville, Illinois
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - Buynak Clinical Research, Valparaiso, Indiana
  - Phoenix Medical Research, Inc., Prairie Village, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Lake Charles Clinical Trials, LLC, Lake Charles, Louisiana
  - Pharmasite Research, Inc., Baltimore, Maryland
  - Potomac Grove Clinical Research Center, Gaithersburg, Maryland
  - Boston Clinical Trials & Medical Research, Boston, Massachusetts
  - Univ. of Massachussetts Memorial Health Care Systems, Worcester, Massachusetts
  - Altea Research Institute, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Erie County Medical Center Corporation, Buffalo, New York
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - CNS Research Science, Inc., Jamaica, New York
  - Village Clinical Research, Inc., New York, New York
  - Manhattan Behavioral Medicine, PLLC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Montefiore Medical Center PRIME, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Clinical Trials of America, Inc, Hickory, North Carolina
  - NorthCoast Clinical Trials, Inc., Beachwood, Ohio
  - Patient Priority Clinical Sites, LLC, Cincinnati, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Inc., Oklahoma City, Oklahoma
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc., Portland, Oregon
  - Suburban Research Associates, Media, Pennsylvania
  - Keystone Clinical Studies, LLC, Norristown, Pennsylvania
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - Lincoln Research, Lincoln, Rhode Island
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Coastal Carolina Research Center, Inc, Mt. Pleasant, South Carolina
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - FutureSearch Clinical Trials, L.P., Austin, Texas
  - BioBehavioral Research of Austin, Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Bayou City Research, Ltd., Houston, Texas
  - Houston Clinical Trials, LLC, Houston, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Radiant Research, Inc., Murray, Utah
  - Neuropsychiatric Associates, Woodstock, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Eastside Therapeutic Resource, Everett, Washington
  - Summit Research Network (Seattle), LLC, Seattle, Washington
  - Frontier Institute, Spokane, Washington
  - Northbrooke Research Center, Brown Deer, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Thase ME, Jacobsen PL, Hanson E, Xu R, Tolkoff M, Murthy NV. Vortioxetine 5, 10, and 20 mg significantly reduces the risk of relapse compared with placebo in patients with remitted major depressive disorder: The RESET study. J Affect Disord. 2022 Apr 15;303:123-130. doi: 10.1016/j.jad.2022.02.002. Epub 2022 Feb 5. PMID 35131363

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 74 investigative sites in the United States from 10 February 2015 to 25 April 2019.
Pre-assignment Details: Participants with diagnosis of major depressive disorder (MDD) were enrolled to receive vortioxetine 10 mg in the Open-label Period for up to 16 weeks. Responders (defined below) were randomized in 1:1:1:1 ratio to receive vortioxetine 5 mg, 10 mg or 20 mg or placebo for up to 32 weeks in the Double-blind Period.
Period: Open-label Period
Arm/Group | Open-label: Vortioxetine 10 mg | Double-blind: Placebo | Double-blind: Vortioxetine 5 mg | Double-blind: Vortioxetine 10 mg | Double-blind: Vortioxetine 20 mg
Started | 1106 | 0 | 0 | 0 | 0
Completed | 580 | 0 | 0 | 0 | 0
Not Completed | 526 | 0 | 0 | 0 | 0
Not completed — Pretreatment Event/Adverse Event | 63 | 0 | 0 | 0 | 0
Not completed — Significant Protocol Deviation | 19 | 0 | 0 | 0 | 0
Not completed — Noncompliance with Study Drug | 10 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 55 | 0 | 0 | 0 | 0
Not completed — Voluntary Withdrawal | 91 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 116 | 0 | 0 | 0 | 0
Not completed — Did not Meet Randomization Criteria | 162 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 9 | 0 | 0 | 0 | 0
Period: Double-blind Period
Arm/Group | Open-label: Vortioxetine 10 mg | Double-blind: Placebo | Double-blind: Vortioxetine 5 mg | Double-blind: Vortioxetine 10 mg | Double-blind: Vortioxetine 20 mg
Started | 0 | 151 | 140 | 145 | 144
Completed | 0 | 70 | 84 | 96 | 86
Not Completed | 0 | 81 | 56 | 49 | 58
Not completed — Pretreatment Event/Adverse Event | 0 | 4 | 3 | 2 | 9
Not completed — Significant Protocol Deviation | 0 | 2 | 7 | 3 | 3
Not completed — Noncompliance with Study Drug | 0 | 1 | 2 | 2 | 3
Not completed — Lost to Follow-up | 0 | 8 | 8 | 6 | 5
Not completed — Voluntary Withdrawal | 0 | 12 | 8 | 9 | 11
Not completed — Relapse | 0 | 50 | 25 | 25 | 26
Not completed — Reason not Specified | 0 | 3 | 3 | 2 | 1
Not completed — Missing | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set for Open-label Period included all participant who received at least 1 dose of Open-label study medication. Baseline I is defined as the last non-missing observation prior to the first dose of open-label study drug.
Arm/Group | Open-label: Vortioxetine 10 mg
Number analyzed (Participants) | 1106
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 807
  Male | 299
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 145
  Not Hispanic or Latino | 961
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7
  Asian | 19
  Native Hawaiian or Other Pacific Islander | 10
  Black or African American | 258
  White | 790
  More than one race | 19
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1106
Height [Mean (Standard Deviation); unit: cm] | 167.7 (9.38)
Weight [Mean (Standard Deviation); unit: kg] | 82.92 (18.695)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=Weight (kg)/height (m^2)
  kg/m^2 | 29.39 (5.731)
Smoking Classification [Count of Participants; unit: Participants]
  Participant has Never Smoked | 705
  Participant is a Current Smoker | 215
  Participant is an Ex-smoker | 186
Alcohol Consumption [Count of Participants; unit: Participants]
  Participant has Never Consumed | 332
  Consumes Once Monthly or Less Consumes Often | 286
  Consumes Once a Week | 167
  Consumes 2 to 6 Times per Week | 159
  Consumes Daily | 11
  Participant was an Ex-Drinker | 151

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to Relapse of Major Depressive Disorder During the First 28 Weeks of the 32-Week Double-Blind Treatment Period
Description: Relapse was defined as either 1) MADRS Score ≥22, 2) lack of efficacy as determined by the investigator or 3) other unsatisfactory treatment response judged by the investigator. Time to relapse was defined as date of relapse - date of randomization + 1 (where date of relapse is the date of last dose, or date of last contact if date of last dose is missing, for participant with a relapse). Participants without relapse were censored at date of withdrawal or date of Week 28 visit, whichever was earliest. MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (i.e., apparent sadness, reported sadness, inner tension, etc.) rated on a 7-point Likert scale from 0 (normal) to 6 (most abnormal) with a total score ranges from 0 to 60. Higher scores indicate greater severity of symptoms. The inter-quartile range (IQR) was 25th percentile to 75th percentile.
Time Frame: From date of double-blind randomization (Week 16) up to relapse or first 28 weeks of Double-blind Period which occurs first (Up to Week 44)
Population: Full Analysis Set (FAS) included all participants who were randomized in the double-blind period and received at least 1 dose of double-blind study drug.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Double-blind: Placebo | Double-blind: Vortioxetine 5 mg | Double-blind: Vortioxetine 10 mg | Double-blind: Vortioxetine 20 mg
Number analyzed (Participants) | 151 | 140 | 145 | 144
weeks | NA [12 to NA] — Median and upper limit of IQR were not reached due to low number of participants with events. | NA [28 to NA] — Median and upper limit of IQR were not reached due to low number of participants with events. | NA [28 to NA] — Median and upper limit of IQR were not reached due to low number of participants with events. | NA [28 to NA] — Median and upper limit of IQR were not reached due to low number of participants with events.
Statistical Analysis 1: Comparison: Double-blind: Vortioxetine 5 mg; Double-blind Vortioxetine 5mg Vs Double-blind Placebo; Test type: Superiority; p = 0.006, Cox Proportional Hazards Model — Gate-keeping fixed-sequence testing procedure was used for multiple comparisons; Cox proportional hazards model with a factor for treatment and baseline II MADRS total score as a covariate, using the exact method to handle ties; Hazard Ratio (HR) = 0.517, 95% CI 2-sided [0.323 to 0.828]
Statistical Analysis 2: Comparison: Double-blind: Vortioxetine 10 mg; Double-blind Vortioxetine 10 mg Vs Double-blind Placebo; Test type: Superiority; p = 0.002, Cox Proportional Hazards Model — Gate-keeping fixed-sequence testing procedure was used for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.476, 95% CI 2-sided [0.296 to 0.767]
Statistical Analysis 3: Comparison: Double-blind: Vortioxetine 20 mg; Double-blind Vortioxetine 20 mg Vs Double-blind Placebo; Test type: Superiority; p = 0.003, Cox Proportional Hazards Model — Gate-keeping fixed-sequence testing procedure was used for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.483, 95% CI 2-sided [0.298 to 0.782]

2. Secondary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (i.e., apparent sadness, reported sadness, inner tension, etc.) rated on a 7-point Likert scale from 0 (normal) to 6 (most abnormal) with a total score range from 0 to 60. Higher score indicates greater severity of symptoms. Baseline II is defined as the last non-missing observation prior to the first dose of double-blind study drug. Mixed model for repeated measures (MMRM) was used for analyses.
Time Frame: Double-blind Baseline (BL) II and Double-blind Period: Weeks 2, 4, 8, 12, 16, 20, 24, 28, and 32
Population: FAS included all participants who were randomized in the double-blind period and received at least 1 dose of double-blind study drug. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Double-blind: Placebo | Double-blind: Vortioxetine 5 mg | Double-blind: Vortioxetine 10 mg | Double-blind: Vortioxetine 20 mg
Number analyzed (Participants) | 151 | 140 | 145 | 144
scores on scale
  Change From BL II at Week 2: number analyzed (Participants) | 148 | 138 | 144 | 140
  Change From BL II at Week 2 | 2.70 (0.461) | 2.23 (0.490) | 1.47 (0.471) | 2.29 (0.481)
  Change From BL II at Week 4: number analyzed (Participants) | 136 | 132 | 137 | 125
  Change From BL II at Week 4 | 4.99 (0.576) | 2.56 (0.599) | 1.98 (0.581) | 2.48 (0.602)
  Change From BL II at Week 8: number analyzed (Participants) | 121 | 123 | 128 | 116
  Change From BL II at Week 8 | 5.98 (0.688) | 3.03 (0.698) | 2.14 (0.679) | 2.97 (0.708)
  Change From BL II at Week 12: number analyzed (Participants) | 104 | 114 | 117 | 110
  Change From BL II at Week 12 | 6.43 (0.704) | 3.51 (0.701) | 1.92 (0.684) | 2.79 (0.707)
  Change From BL II at Week 16: number analyzed (Participants) | 90 | 108 | 113 | 105
  Change From BL II at Week 16 | 5.77 (0.724) | 3.73 (0.707) | 2.08 (0.688) | 3.14 (0.712)
  Change From BL II at Week 20: number analyzed (Participants) | 83 | 102 | 107 | 100
  Change From BL II at Week 20 | 5.95 (0.699) | 3.34 (0.673) | 1.86 (0.653) | 3.18 (0.675)
  Change From BL II at Week 24: number analyzed (Participants) | 78 | 95 | 103 | 97
  Change From BL II at Week 24 | 5.69 (0.765) | 3.78 (0.733) | 2.19 (0.707) | 3.16 (0.730)
  Change From BL II at Week 28: number analyzed (Participants) | 71 | 90 | 100 | 91
  Change From BL II at Week 28 | 5.07 (0.774) | 3.18 (0.730) | 2.72 (0.699) | 3.20 (0.726)
  Change From BL II at Week 32: number analyzed (Participants) | 67 | 85 | 94 | 87
  Change From BL II at Week 32 | 6.55 (0.858) | 3.46 (0.815) | 2.58 (0.784) | 2.97 (0.815)
Statistical Analysis 1: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Change From Baseline II at Week 2; Test type: Superiority; p = 0.421, MMRM; MMRM with treatment, visit, BL II score, treatment by visit interaction as fixed factors, center as random effect, and unstructured covariance matrix; Least Squares Mean (LSM) Difference = -0.48, 95% CI 2-sided [-1.63 to 0.68], Standard Error of Mean 0.590
Statistical Analysis 2: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Change From Baseline II at Week 2; Test type: Superiority; p = 0.037, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.23, 95% CI 2-sided [-2.39 to -0.08], Standard Error of Mean 0.589
Statistical Analysis 3: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Change From Baseline II at Week 2; Test type: Superiority; p = 0.488, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.41, 95% CI 2-sided [-1.57 to 0.75], Standard Error of Mean 0.592
Statistical Analysis 4: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Change From Baseline II at Week 4; Test type: Superiority; p = 0.002, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.43, 95% CI 2-sided [-3.93 to -0.93], Standard Error of Mean 0.765
Statistical Analysis 5: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Change From Baseline II at Week 4; Test type: Superiority; p < 0.001, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.00, 95% CI 2-sided [-4.49 to -1.51], Standard Error of Mean 0.761
Statistical Analysis 6: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Change From Baseline II at Week 4; Test type: Superiority; p = 0.001, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.50, 95% CI 2-sided [-4.02 to -0.98], Standard Error of Mean 0.775
Statistical Analysis 7: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Change From Baseline II at Week 8; Test type: Superiority; p = 0.001, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.95, 95% CI 2-sided [-4.76 to -1.13], Standard Error of Mean 0.924
Statistical Analysis 8: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Change From Baseline II at Week 8; Test type: Superiority; p < 0.001, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.84, 95% CI 2-sided [-5.64 to -2.03], Standard Error of Mean 0.919
Statistical Analysis 9: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Change From Baseline II at Week 8; Test type: Superiority; p = 0.001, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.00, 95% CI 2-sided [-4.84 to -1.16], Standard Error of Mean 0.939
Statistical Analysis 10: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Change From Baseline II at Week 12; Test type: Superiority; p = 0.002, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.92, 95% CI 2-sided [-4.76 to -1.08], Standard Error of Mean 0.938
Statistical Analysis 11: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Change From Baseline II at Week 12; Test type: Superiority; p < 0.001, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.51, 95% CI 2-sided [-6.34 to -2.68], Standard Error of Mean 0.934
Statistical Analysis 12: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Change From Baseline II at Week 12; Test type: Superiority; p < 0.001, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.64, 95% CI 2-sided [-5.50 to -1.78], Standard Error of Mean 0.949
Statistical Analysis 13: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Change From Baseline II at Week 16; Test type: Superiority; p = 0.033, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.04, 95% CI 2-sided [-3.92 to -0.16], Standard Error of Mean 0.957
Statistical Analysis 14: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Change From Baseline II at Week 16; Test type: Superiority; p < 0.001, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.69, 95% CI 2-sided [-5.55 to -1.82], Standard Error of Mean 0.952
Statistical Analysis 15: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Change From Baseline II at Week 16; Test type: Superiority; p = 0.007, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.63, 95% CI 2-sided [-4.52 to -0.73], Standard Error of Mean 0.967
Statistical Analysis 16: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Change From Baseline II at Week 20; Test type: Superiority; p = 0.004, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.61, 95% CI 2-sided [-4.40 to -0.82], Standard Error of Mean 0.912
Statistical Analysis 17: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Change From Baseline II at Week 20; Test type: Superiority; p < 0.001, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.09, 95% CI 2-sided [-5.86 to -2.31], Standard Error of Mean 0.906
Statistical Analysis 18: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Change From Baseline II at Week 20; Test type: Superiority; p = 0.003, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.76, 95% CI 2-sided [-4.57 to -0.96], Standard Error of Mean 0.921
Statistical Analysis 19: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Change From Baseline II at Week 24; Test type: Superiority; p = 0.057, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.92, 95% CI 2-sided [-3.89 to 0.06], Standard Error of Mean 1.008
Statistical Analysis 20: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Change From Baseline II at Week 24; Test type: Superiority; p < 0.001, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.50, 95% CI 2-sided [-5.46 to -1.55], Standard Error of Mean 0.997
Statistical Analysis 21: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Change From Baseline II at Week 24; Test type: Superiority; p = 0.012, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.53, 95% CI 2-sided [-4.51 to -0.55], Standard Error of Mean 1.011
Statistical Analysis 22: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Change From Baseline II at Week 28; Test type: Superiority; p = 0.061, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.90, 95% CI 2-sided [-3.88 to 0.09], Standard Error of Mean 1.012
Statistical Analysis 23: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Change From Baseline II at Week 28; Test type: Superiority; p = 0.018, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.36, 95% CI 2-sided [-4.31 to -0.40], Standard Error of Mean 0.997
Statistical Analysis 24: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Change From Baseline II at Week 28; Test type: Superiority; p = 0.065, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.88, 95% CI 2-sided [-3.87 to 0.12], Standard Error of Mean 1.015
Statistical Analysis 25: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Change From Baseline II at Week 32; Test type: Superiority; p = 0.007, MMRM; [statistical method as in outcome 2, analysis 1]; MMRM Model = -3.09, 95% CI 2-sided [-5.31 to -0.86], Standard Error of Mean 1.136
Statistical Analysis 26: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Change From Baseline II at Week 32; Test type: Superiority; p < 0.001, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.97, 95% CI 2-sided [-6.16 to -1.77], Standard Error of Mean 1.122
Statistical Analysis 27: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Change From Baseline II at Week 32; Test type: Superiority; p = 0.002, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.58, 95% CI 2-sided [-5.82 to -1.34], Standard Error of Mean 1.143

3. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale-Severity (CGI-S) Score at Each Week Assessed
Description: The CGI-S is a 7-point scale that requires the clinician to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with participant who have the same diagnosis. Considering total clinical experience, a participant was assessed on severity of mental illness on the following scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=extremely ill. Baseline II is defined as the last non-missing observation prior to the first dose of double-blind study drug. MMRM was used for analyses.
Time Frame: Double-blind Baseline (BL) II and Double-blind Period: Weeks 2, 4, 8, 12, 16, 20, 24, 28, and 32
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Double-blind: Placebo | Double-blind: Vortioxetine 5 mg | Double-blind: Vortioxetine 10 mg | Double-blind: Vortioxetine 20 mg
Number analyzed (Participants) | 151 | 140 | 145 | 144
scores on scale
  Change From BL II at Week 2: number analyzed (Participants) | 147 | 138 | 144 | 140
  Change From BL II at Week 2 | 0.35 (0.065) | 0.32 (0.069) | 0.26 (0.067) | 0.27 (0.068)
  Change From BL II at Week 4: number analyzed (Participants) | 135 | 132 | 135 | 125
  Change From BL II at Week 4 | 0.61 (0.075) | 0.32 (0.078) | 0.30 (0.076) | 0.25 (0.078)
  Change From BL II at Week 8: number analyzed (Participants) | 121 | 122 | 127 | 115
  Change From BL II at Week 8 | 0.68 (0.091) | 0.38 (0.092) | 0.29 (0.089) | 0.30 (0.093)
  Change From BL II at Week 12: number analyzed (Participants) | 104 | 113 | 116 | 109
  Change From BL II at Week 12 | 0.74 (0.092) | 0.46 (0.091) | 0.24 (0.089) | 0.35 (0.092)
  Change From BL II at Week 16: number analyzed (Participants) | 90 | 107 | 113 | 104
  Change From BL II at Week 16 | 0.62 (0.094) | 0.50 (0.091) | 0.25 (0.088) | 0.34 (0.091)
  Change From BL II at Week 20: number analyzed (Participants) | 83 | 102 | 107 | 100
  Change From BL II at Week 20 | 0.61 (0.094) | 0.40 (0.089) | 0.17 (0.086) | 0.28 (0.089)
  Change From BL II at Week 24: number analyzed (Participants) | 77 | 94 | 103 | 97
  Change From BL II at Week 24 | 0.60 (0.103) | 0.45 (0.098) | 0.24 (0.094) | 0.37 (0.097)
  Change From BL II at Week 28: number analyzed (Participants) | 70 | 89 | 100 | 91
  Change From BL II at Week 28 | 0.45 (0.101) | 0.33 (0.094) | 0.30 (0.090) | 0.34 (0.093)
  Change From BL II at Week 32: number analyzed (Participants) | 66 | 85 | 94 | 87
  Change From BL II at Week 32 | 0.59 (0.108) | 0.41 (0.101) | 0.26 (0.097) | 0.22 (0.100)
Statistical Analysis 1: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Change From Baseline II at Week 2; Test type: Superiority; p = 0.732, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.03, 95% CI 2-sided [-0.20 to 0.14], Standard Error of Mean 0.085
Statistical Analysis 2: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Change From Baseline II at Week 2; Test type: Superiority; p = 0.273, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.09, 95% CI 2-sided [-0.26 to 0.07], Standard Error of Mean 0.085
Statistical Analysis 3: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Change From Baseline II at Week 2; Test type: Superiority; p = 0.361, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.08, 95% CI 2-sided [-0.24 to 0.09], Standard Error of Mean 0.085
Statistical Analysis 4: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Change From Baseline II at Week 4; Test type: Superiority; p = 0.004, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.28, 95% CI 2-sided [-0.48 to -0.09], Standard Error of Mean 0.099
Statistical Analysis 5: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Change From Baseline II at Week 4; Test type: Superiority; p = 0.002, Least Squares Mean Difference; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.31, 95% CI 2-sided [-0.50 to -0.12], Standard Error of Mean 0.099
Statistical Analysis 6: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Change From Baseline II at Week 4; Test type: Superiority; p < 0.001, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.36, 95% CI 2-sided [-0.55 to -0.16], Standard Error of Mean 0.100
Statistical Analysis 7: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Change From Baseline II at Week 8; Test type: Superiority; p = 0.014, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.30, 95% CI 2-sided [-0.54 to -0.06], Standard Error of Mean 0.121
Statistical Analysis 8: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Change From Baseline II at Week 8; Test type: Superiority; p = 0.001, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.39, 95% CI 2-sided [-0.63 to -0.16], Standard Error of Mean 0.121
Statistical Analysis 9: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Change From Baseline II at Week 8; Test type: Superiority; p = 0.002, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.38, 95% CI 2-sided [-0.62 to -0.14], Standard Error of Mean 0.123
Statistical Analysis 10: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Change From Baseline II at Week 12; Test type: Superiority; p = 0.025, Least Squares Mean Difference; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.27, 95% CI 2-sided [-0.51 to -0.03], Standard Error of Mean 0.122
Statistical Analysis 11: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Change From Baseline II at Week 12; Test type: Superiority; p < 0.001, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.50, 95% CI 2-sided [-0.74 to -0.26], Standard Error of Mean 0.122
Statistical Analysis 12: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Change From Baseline II at Week 12; Test type: Superiority; p = 0.002, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.39, 95% CI 2-sided [-0.63 to -0.15], Standard Error of Mean 0.124
Statistical Analysis 13: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Change From Baseline II at Week 16; Test type: Superiority; p = 0.333, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.12, 95% CI 2-sided [-0.36 to 0.12], Standard Error of Mean 0.123
Statistical Analysis 14: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Change From Baseline II at Week 16; Test type: Superiority; p = 0.002, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.37, 95% CI 2-sided [-0.61 to -0.13], Standard Error of Mean 0.122
Statistical Analysis 15: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Change From Baseline II at Week 16; Test type: Superiority; p = 0.023, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.28, 95% CI 2-sided [-0.53 to -0.04], Standard Error of Mean 0.124
Statistical Analysis 16: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Change From Baseline II at Week 20; Test type: Superiority; p = 0.092, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.20, 95% CI 2-sided [-0.44 to 0.03], Standard Error of Mean 0.121
Statistical Analysis 17: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Change From Baseline II at Week 20; Test type: Superiority; p < 0.001, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.44, 95% CI 2-sided [-0.67 to -0.20], Standard Error of Mean 0.121
Statistical Analysis 18: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Change From Baseline II at Week 20; Test type: Superiority; p = 0.008, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.33, 95% CI 2-sided [-0.57 to -0.09], Standard Error of Mean 0.122
Statistical Analysis 19: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Change From Baseline II at Week 24; Test type: Superiority; p = 0.248, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.16, 95% CI 2-sided [-0.42 to 0.11], Standard Error of Mean 0.135
Statistical Analysis 20: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Change From Baseline II at Week 24; Test type: Superiority; p = 0.006, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.37, 95% CI 2-sided [-0.63 to -0.10], Standard Error of Mean 0.133
Statistical Analysis 21: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Change From Baseline II at Week 24; Test type: Superiority; p = 0.087, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.23, 95% CI 2-sided [-0.50 to 0.03], Standard Error of Mean 0.135
Statistical Analysis 22: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Change From Baseline II at Week 28; Test type: Superiority; p = 0.362, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.12, 95% CI 2-sided [-0.38 to 0.14], Standard Error of Mean 0.131
Statistical Analysis 23: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Change From Baseline II at Week 28; Test type: Superiority; p = 0.251, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.15, 95% CI 2-sided [-0.40 to 0.10], Standard Error of Mean 0.129
Statistical Analysis 24: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Change From Baseline II at Week 28; Test type: Superiority; p = 0.391, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.11, 95% CI 2-sided [-0.37 to 0.14], Standard Error of Mean 0.131
Statistical Analysis 25: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Change From Baseline II at Week 32; Test type: Superiority; p = 0.209, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.18, 95% CI 2-sided [-0.45 to 0.10], Standard Error of Mean 0.141
Statistical Analysis 26: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Change From Baseline II at Week 32; Test type: Superiority; p = 0.018, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.33, 95% CI 2-sided [-0.60 to -0.06], Standard Error of Mean 0.139
Statistical Analysis 27: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Change From Baseline II at Week 32; Test type: Superiority; p = 0.009, MMRM; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.37, 95% CI 2-sided [-0.65 to -0.09], Standard Error of Mean 0.141

4. Secondary Outcome: Clinical Global Impression Scale-Global Improvement Scale (CGI-I) Score
Description: The CGI-I scale assesses the participant's improvement (or worsening) as assessed by the clinician relative to Baseline on a 7-point scale where 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse.
Time Frame: Week 32
Population: FAS included all participants who were randomized in the double-blind period and received at least 1 dose of double-blind study drug. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Double-blind: Placebo | Double-blind: Vortioxetine 5 mg | Double-blind: Vortioxetine 10 mg | Double-blind: Vortioxetine 20 mg
Number analyzed (Participants) | 119 | 120 | 126 | 144
scores on scale | 4.4 (1.47) | 3.9 (1.51) | 3.5 (1.72) | 3.7 (1.56)

5. Secondary Outcome: Time From Randomization to Relapse of Major Depressive Disorder During the Entire 32-Week Double-Blind Treatment Period
Description: Relapse was defined as either 1) MADRS Score ≥22, 2) lack of efficacy as determined by the investigator or 3) other unsatisfactory treatment response judged by the investigator. Time to relapse was defined as date of relapse - date of randomization + 1 (where date of relapse is the date of last dose, or date of last contact if date of last dose is missing, for participant with a relapse). Participants without relapse were censored. MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (i.e., apparent sadness, reported sadness, inner tension, etc.) rated on a 7-point Likert scale from 0 (normal) to 6 (most abnormal) with a total score ranges from 0 to 60. Higher scores indicate greater severity of symptoms. The IQR was 25th percentile to 75th percentile.
Time Frame: From date of double-blind randomization (Week 16) up to relapse or 32 weeks of Double-blind Period which occurs first (Up to Week 44)
Population: FAS included all participants who were randomized in the double-blind period and received at least 1 dose of double-blind study drug.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Double-blind: Placebo | Double-blind: Vortioxetine 5 mg | Double-blind: Vortioxetine 10 mg | Double-blind: Vortioxetine 20 mg
Number analyzed (Participants) | 151 | 140 | 145 | 144
weeks | NA [12 to NA] — Median and upper limit of IQR was not reached due to low number of participants with events. | NA [32 to NA] — Median and upper limit of IQR was not reached due to low number of participants with events. | NA [32 to NA] — Median and upper limit of IQR was not reached due to low number of participants with events. | NA [32 to NA] — Median and upper limit of IQR was not reached due to low number of participants with events.
Statistical Analysis 1: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 5 mg; Double-blind Vortioxetine 5mg Vs Double-blind Placebo; Test type: Superiority; p = 0.002, Cox Proportional Hazards Model — Gate-keeping fixed-sequence testing procedure was used for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.481, 95% CI 2-sided [0.302 to 0.766]
Statistical Analysis 2: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 10 mg; Double-blind Vortioxetine 10 mg Vs Double-blind Placebo; Test type: Superiority; p < 0.001, Cox Proportional Hazards Model — Gate-keeping fixed-sequence testing procedure was used for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.455, 95% CI 2-sided [0.286 to 0.725]
Statistical Analysis 3: Comparison: Double-blind: Placebo vs Double-blind: Vortioxetine 20 mg; Double-blind Vortioxetine 20 mg Vs Double-blind Placebo; Test type: Superiority; p = 0.002, Cox Proportional Hazards Model — Gate-keeping fixed-sequence testing procedure was used for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.484, 95% CI 2-sided [0.304 to 0.771]

ADVERSE EVENTS:
Time Frame: From first dose of study drug and up to 30 days after the last dose (Up to 48 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Open-label: Vortioxetine 10 mg | Double-blind: Placebo | Double-blind: Vortioxetine 5 mg | Double-blind: Vortioxetine 10 mg | Double-blind: Vortioxetine 20 mg
All-Cause Mortality (participants affected / at risk) | 0/1106 | 0/151 | 0/140 | 1/145 | 0/144
Serious Adverse Events (participants affected / at risk) | 9/1106 | 1/151 | 3/140 | 4/145 | 0/144
Other Adverse Events (participants affected / at risk) | 417/1106 | 16/151 | 30/140 | 27/145 | 32/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label: Vortioxetine 10 mg (N=1106) | Double-blind: Placebo (N=151) | Double-blind: Vortioxetine 5 mg (N=140) | Double-blind: Vortioxetine 10 mg (N=145) | Double-blind: Vortioxetine 20 mg (N=144)
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Post procedural cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with vortioxetine 10 mg and was not related.
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label: Vortioxetine 10 mg (N=1106) | Double-blind: Placebo (N=151) | Double-blind: Vortioxetine 5 mg (N=140) | Double-blind: Vortioxetine 10 mg (N=145) | Double-blind: Vortioxetine 20 mg (N=144)
Upper respiratory tract infection (Infections and infestations) | 0 | 6 | 9 | 9 | 9
Nasopharyngitis (Infections and infestations) | 56 | 4 | 7 | 7 | 8
Nausea (Gastrointestinal disorders) | 292 | 2 | 4 | 5 | 13
Weight increased (Investigations) | 0 | 3 | 5 | 7 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 8 | 0 | 2
Headache (Nervous system disorders) | 91 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 58 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT02371980/SAP_000.pdf
  • Study Protocol (2015-09-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT02371980/Prot_001.pdf